CLINICAL TRIAL: NCT00275171
Title: The Effect of 0.1 mg Recombinant Human Thyrotropin (rhTSH) on Thyroid Radioiodine-uptake and the Degree of Goiter Reduction Following 131I-therapy, in Patients With Benign Non-toxic Nodular Goiter. A Randomized, Double-blind, Placebo-controlled Trial.
Brief Title: rhTSH, Radioiodine Uptake and Goiter Reduction Following 131I Therapy in Patients With Benign Nontoxic Nodular Goiter
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Steen Bonnema (Other)
Responsible Party: Sponsor-Investigator, Steen Bonnema, Consultant, phd, DMsc, Odense University Hospital
Organization: Odense University Hospital (Other)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 019
Record Dates: First submitted 2006-01-09; First posted 2006-01-11 (Estimated); Last update posted 2013-12-04 (Estimated); Status verified 2013-12

CONDITIONS: Nodular Goiter
Keywords: Nontoxic nodular goiter; 131I therapy; thyroid radioiodine uptake; optimal time-interval; reduced 131I activity; goiter reduction
MeSH Terms: conditions — Goiter, Nodular | interventions — Thyrotropin Alfa

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- rhTSH (Active Comparator): proceeded by 0.1 mg rhTSH
  Interventions: Drug: Recombinant human thyrotropin (Thyrogen); Drug: recombinant human TSH
- Placebo (Placebo Comparator): 1 ml isotonic saline
  Interventions: Other: isotonic saline = placebo

INTERVENTIONS:
Drug: Recombinant human thyrotropin (Thyrogen) — 0.1 mg rhTSH administered intramuscularly
  Arms: rhTSH
Drug: recombinant human TSH — 0.1 mg rhTSH administered intramuscularly
  Arms: rhTSH
Other: isotonic saline = placebo — 0.1 mg isotonic saline injected intramuscularly
  Arms: Placebo

SUMMARY:
The study aims at clarifying (in a randomized, double-blinded design):

1. Whether stimulation with 0.1 mg rhTSH 24, 48 or 72 hours before induction of a 131I-tracer dosis increases the 131I uptake in patients with atoxic multinodular goitre and to study which time interval is the most optimal (Part I)
2. Whether patients suffering from atoxic multinodular goitre obtains a corresponding goitre reduction compared with a control group when stimulating with 0.1 mg rh TSH 24, 48 or 72 hours before 131I therapy and when reducing the thyroid radiation dose to 50 Gy (Part II)

The two studies will be carried out successively on the same patient population. The 131I uptake will be carried out first followed by the I therapy itself. The patients are compared with a placebo-treated control group going through the same course of treatment, but the 131I dosis will be 100 Gy (standard treatment). After the 131I therapy, all patients are followed during one year with a regular ultrasound scan of the thyroid gland and control of the metabolic status. The patient satisfaction is monitored by the use of a visual-analogue-scale.

ELIGIBILITY:
Inclusion Criteria:

* Age over 18 years
* Apart from benign non-toxic goiter no other serious illness
* Signed proof of participation

Exclusion Criteria:

* Treatment with Levothyroxine
* Former 131I-therapy
* A thyroid volume above 100 ml or a retro-clavicular component
* Unsafe contraception
* Pregnancy or breastfeeding
* Participation in another clinical trial
* Previous allergic reaction toward rhTSH
* Suspicion of malignancy in the thyroid gland either by clinical examination, laboratory findings (a raised serum calcitonin or ionized calcium)or by fine-needle aspiration biopsy
* Physically or mental condition making it impossible to participate
* Acute ischemic heart attach within the last 3 months
* Alcohol and/or drug addicts

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 90 (Actual)
Dates: Start 2006-02; Primary Completion 2009-04 (Actual); Study Completion 2009-09 (Actual)

PRIMARY OUTCOMES:
An intra-individual comparison of the thyroid 131I-uptake before and after stimulation with rhTSH /placebo | 24 and 96 hours after tracer administration
An inter-individual comparison of the thyroid 131I uptake between those who receive placebo and those who receive rhTSH | 24 and 96 hours after tracer administration
An estimation of which time-interval, injecting rhTSH, that is more favourable before 131I therapy (24 hours, 48 hours or 72 hours) | 24 and 96 hours after tracer administration
A comparison of the degree of goiter reduction when patients are prestimulated with rhTSH and receive a thyroid 131I dose of 50 Gy or when receiving conventional 131I, receiving a thyroid dose of 100 Gy | 3, 6, 9 and 12 months after 131I therapy

SECONDARY OUTCOMES:
A registration of adverse effects following rhTSH/placebo | All adverse effects occuring within one year follow-up
Patient satisfaction (Visual Analogue Scale) before, 3 months post 131I therapy, and at the end of follow-up (1 year). | baseline, 3 and 12 months after 131I therapy
Development of TPOab or TSHRab | At 12 months follow-up
Thyroid function | At 12 months follow up.

CONTACTS AND LOCATIONS:
Overall Officials: Steen J. Bonnema, MD, Principal Investigator — Odense University Hospital
Locations (1):
- Odense University Hospital, Odense, Denmark

REFERENCES:
- [Derived] Huo Y, Xie J, Chen S, Wang H, Ma C. Recombinant human thyrotropin (rhTSH)-aided radioiodine treatment for non-toxic multinodular goitre. Cochrane Database Syst Rev. 2021 Dec 28;12(12):CD010622. doi: 10.1002/14651858.CD010622.pub2. PMID 34961921
- [Derived] Fast S, Hegedus L, Grupe P, Nielsen VE, Bluhme C, Bastholt L, Bonnema SJ. Recombinant human thyrotropin-stimulated radioiodine therapy of nodular goiter allows major reduction of the radiation burden with retained efficacy. J Clin Endocrinol Metab. 2010 Aug;95(8):3719-25. doi: 10.1210/jc.2010-0634. Epub 2010 Jun 2. PMID 20519346